CLINICAL TRIAL: NCT02538653
Title: Determination of the Postprandial Responses to Two Cereal Foods Differing by Their SDS Content Consumed Alone.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KBE042
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Metabolic Disorder; Carbohydrate, Absorption, Intestine
Keywords: glycemic & insulin response, SDS, cereal product, Nutrition
MeSH Terms: conditions — Metabolic Diseases; Shwachman-Diamond Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sandwich biscuits high in SDS (Experimental): 50 g of sandwich product with high level of SDS together with a glass of 250 mL of Evian water.
  Interventions: Other: Sandwich biscuit high in SDS
- Co-extruded cereals low in SDS (Active Comparator): 48.3 g of co-extruded cereals low in SDS together with a glass of 250 mL of Evian water.
  Interventions: Other: Co-extruded cereal low in SDS

INTERVENTIONS:
Other: Sandwich biscuit high in SDS — Consumption of the high SDS product (50g) alone with a glass of water
  Arms: Sandwich biscuits high in SDS
Other: Co-extruded cereal low in SDS — Consumption of the low SDS product (48.3 g) alone with a glass of water
  Arms: Co-extruded cereals low in SDS

SUMMARY:
This study aimed at determining the 4-hours postprandial blood glucose and insulin responses to the ingestion of cereal product differing by their SDS content.

DETAILED DESCRIPTION:
This study aimed at determining the 4-hours postprandial blood glucose and insulin responses to the ingestion of cereal product differing by their SDS content. It is a laboratory-based research study with an open cross-over design, including 20 healthy non-smoking voluntary subjects, aged from 18 to 45 years. 2 test sessions per subject are included in the study. Foods are consumed in a random order according to a randomisation list.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-45 years.
* Non-smoker.
* BMI values between 19-30 kg/m2 (bounds included). Around half of the subjects will be normal weight and the other half overweight.
* Ethnicity. Subjects should have the closest characteristics compared to the American population. Not less than 75% but not more than 90% of the subjects should be Caucasian. Not more than 10% of the subjects will be of Asian or Asian Indian descent. The remaining subjects will be from other ethnic groups except from Australian Aborigines.
* Healthy subjects with:

  * Normal glucose tolerance (fasting blood glucose < 6.0 mmol/L during the first test session and results of oral glucose tolerance test conducted within the last 30 days within recommendations (fasting blood glucose < 6.0 mmol/L, 120 minute glucose < 8.9 mmol/L))
  * Normal laboratory values for various measures of metabolic health (full blood count, gamma-GT, AST, ALT, glucose, TAGs, total cholesterol, HDL-cholesterol, LDL-cholesterol);
  * Normal systolic blood pressure (100-150 mmHg);
  * Normal diastolic blood pressure (60-90 mmHg);
  * Normal resting heart rate (50-90 beats per minutes after 3 minutes rest).
* Stable dietary habits; normal eating patterns; no history of eating disorders or strict dieting.
* Moderate level of physical activity (from basic daily activity to a high level of physical activity (regular physical activity at least 3 times per week)
* Able to fast for at least 10 hours the night before each test session
* Able to refrain from eating legumes and drinking alcohol the day before each test session.
* Subject covered by social security or covered by a similar system
* Subject not taking any treatment for anorexia, weight loss, or any form of treatment likely tointerfere with metabolism or dietary habits
* Subject having given written consent to take part in the study.

Exclusion Criteria:

* Following a restrictive diet.
* Family history of Diabetes Mellitus or obesity
* Suffering from any clinical, physical or mental illness.
* Suffering from any food allergies or hypersensitivities (wheat, milk, egg, nuts, etc).
* Taking any regular prescription medication at the time of inclusion (except regular oral contraception medication)
* Subject from the Australian Aboriginal ethnicity.
* Female who is pregnant (positive test results), lactating, planning pregnancy or not using acceptable contraceptive.
* Females who consistently suffer from premenstrual tension and marked changes in appetite during their menstrual cycle.
* Subject having taken part in another clinical trial within the last week.
* Subject currently taking part in another clinical trial or being in the exclusion period of another clinical trial.
* Subject undergoing general anaesthesia in the month prior to inclusion.
* Subject in a situation which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Postprandial changes in plasma glucose levels over 2 hours (iAUC [0-120 min]) after consumption of the test products | 2 hours after food consumption

SECONDARY OUTCOMES:
Postprandial changes in glycaemia over 3 hours (iAUC [0-180]), 4h (iAUC[0-240]), during the second part of the morning (iAUC [120-240] and iAUC[180-240]) following the intake of the test products will be analysed. | 4 hours after food consumption
Postprandial changes in insulinemia over 2 hours (iAUC [0-120]), over 3 hours (iAUC [0-180]), 4 hours (iAUC[0-240]), during the second part of the morning (iAUC [120-240] and iAUC [180-240]) following the intake of the test products will be analysed. | 4 hours after food consumption

OTHER OUTCOMES:
The plasma glucose peak value and the time for this latter will also be calculated. | 4 hours after food consumption
The plasma insulin peak value and the time for this latter will also be calculated. | 4 hours after food consumption

CONTACTS AND LOCATIONS:
Overall Officials: Jennie Brand Miller, Principal Investigator — University of Sydney
Locations (1):
- University of Sydney, Sydney, New South Wales, Australia